CLINICAL TRIAL: NCT05154539
Title: Innovation of Hearing Rehabilitation and Effects of Reform
Acronym: InHEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Lene Dahl Siggaard, Principal Investigator, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: InHEAR
Record Dates: First submitted 2021-11-14; First posted 2021-12-13 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: 1:1:1 three arm randomized, controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Group 1 (TG1) (Experimental): TG1 participants are testing the new digital assessment routine in a private setting.
  Audiology assistants in private hearing clinics located in the Region of Northern Jutland in Denmark are performing the standardized examination packages. The private hearing clinics also conduct hearing aid treatment for TG1 participants with simple hearing loss.
  TG21 participants with complicated hearing loss or ear-related diseases are referred to the Department of Audiology at Aalborg University Hospital for further examination prior to treatment initiation.
  Interventions: Diagnostic Test: Remote digital assessment
- Test Group 2 (TG2) (Experimental): TG2 participants are testing the new digital assessment routine in a public setting.
  Audiology assistants in public hearing clinics located in the Region of Northern Jutland in Denmark are performing the standardized examination packages. The public hearing clinics also conduct hearing aid treatment for TG2 participants with simple hearing loss.
  TG2 participants with complicated hearing loss or ear-related diseases are referred to the Department of Audiology at Aalborg University Hospital for further examination prior to treatment initiation.
  Interventions: Diagnostic Test: Remote digital assessment
- Control Group 3 (CG3) (Active Comparator): CG3 participants will be assessed conventionally by a private practicing ENT specialist in the Region of Northern Jutland in Denmark at physical consultation in accordance with current Danish practice. CG3 participants with simple hearing loss can choose whether hearing aid treatment should be conducted in either a private or a public hearing clinic.
  CG3 participants with complicated hearing loss or ear-related diseases are referred to the Department of Audiology at Aalborg University Hospital for further examination prior to treatment initiation.
  Interventions: Diagnostic Test: Conventional physical assessment

INTERVENTIONS:
Diagnostic Test: Remote digital assessment — Remote digital assessment of test group participants
  Arms: Test Group 1 (TG1); Test Group 2 (TG2)
Diagnostic Test: Conventional physical assessment — Conventional physical assessment of control group participants
  Arms: Control Group 3 (CG3)

SUMMARY:
The Danish health care system has been criticized for its structural inefficiency and latency to initiate proper hearing rehabilitation amongst hearing-impaired individuals. Waiting lists are extensive, and audiometries are repeated before hearing aid treatment is initiated. Demographic changes forecast increasing numbers of +65-year-olds and consequently increased demand for hearing rehabilitation. To remedy this situation, the Danish Ministry of Health has proposed a new national initiative to implement innovative digital approaches to improve hearing rehabilitation, including a new, digital remote assessment routine.

The aim of this study is to investigate:

Primarily:

1. Patient safety of remote vs. conventional assessment
2. Patient-reported satisfaction and treatment effect of remote vs. conventional assessment

   Secondarily:
3. Inter-subspecialty and inter-personal assessment differences between four ENT specialists using a remote assessment routine
4. Translation and validation of the Danish adapted version of the Consumer Ear Disease Risk Assessment (CEDRA) questionnaire.

The main study is a randomized clinical trial with three arms and 1:1:1 assignment comprising 751 potential first-time adult hearing aid users.

Since March 2021, 751 patients have been randomized and assigned to 20 different clinics. The remote assessment routine works well for both patients, assessors, and clinics. Inclusion is expected to end in December 2021 and overall study completion is anticipated in april 2022.

Deficient diagnosis of complicating conditions in first time hearing aid users is the main concern in remote assessment. If the study shows the practice to be safe, it could form the foundation of a future nationwide implementation of remote care in Danish hearing rehabilitation.

DETAILED DESCRIPTION:
InHEAR is a prospective randomized controlled trial aimed to investigate a new, Danish digital remote assessment routine applied in 751 hearing-impaired adults. The existing, traditional Danish referral model requires a physical consultation with an ear-nose- and throat (ENT) specialist prior to treatment initiation. The digital referral reform replaces the traditional physical ENT specialist assessment with a standardized examination package performed by educated and experienced audiology assistants, allowing physicians to assess and refer hearing-impaired adults to the relevant treatment regime remotely and asynchronously without meeting the patients physically.

After inclusion, the participants will be randomized equally into three groups:

Test group 1 (TG1) will be testing the digital assessment routine in private hearing clinics.

Test group 2 (TG2) will be testing the digital assessment routine in public hearing clinics.

Control group 3 (CG3) will be assessed in accordance with current Danish practice.

The examination package performed on test group participants comprises of:

1. A standardized, focused medical hearing history record (questionnaire)
2. A standard audiometry test, including air conduction, bone conduction, speech discrimination test and acoustic reflex test
3. Tympanometry
4. Still images of the eardrums performed by video-otoscopy

Four ENT-specialists, two audiologists and to private ENT specialist, will independently and remotely assess the standardized test group examination packages and refer the test group participants to relevant treatment. Participants in the control group are assessed by a private ENT specialist at a physical consultation and referred to relevant treatment in accordance with current Danish practice. Participants with simple hearing loss will be offered hearing rehabilitation with hearing aids. Participants with complicated hearing loss or complicated ear related diseases will be offered a physical ENT specialist assessment at the Department of Audiology at Aalborg University Hospital prior to treatment initiation.

Patient-reported data concerning treatment satisfaction-, quality- and effect will be registered throughout the study period.

Two-three months after treatment initiation, all participants are evaluated by an ENT specialist in Audiology or Otology at a "golden standard" physical consultation at the Department of Audiology at Aalborg University Hospital. Assessment and referral accuracy, patient-reported treatment quality and satisfaction between the test groups and the control group participants will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Subjective hearing difficulty
* Must be able to understand and read Danish

Exclusion Criteria:

* Recent ENT specialist assessment
* Prior HA usage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 751 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis of complicating hearing and/or ear-related conditions in hearing impaired adults | Baseline
  ENT specialist assessments were performed remotely in test group participants and physically in control group participants at baseline. Based on this assessment, participants were divided into three categories of simple hearing loss, severe/complicated hearing loss, and no hearing loss respectively. Hearing aid treatment was administered when indicated.
  The primary focus was to correctly identify participants with severe/complicated hearing loss and/or complicating ear-related conditions in both test and control groups.
Remote ENT specialist assessment: Diagnostic accuracy of severe/complicated hearing loss and/or complicating ear-related conditions in hearing impaired adults. | Month 3
  A physical, "golden standard" ENT assessment was performed in all test group participants after 3 months. Based on this assessment, participants were again divided into categories of simple hearing loss, severe/complicated hearing loss, and no hearing loss respectively. The "golden standard" ENT assessment at Month 3 was compared to the remote ENT assessment at baseline and diagnostic differences were registered.
  Outcome measures: Sensitivity and specificity of the remote ENT specialist assessment routine in identifying severe/complicated hearing loss and/or complicating ear-related conditions in hearing impaired adults.
Conventional, physical ENT specialist assessment: Diagnostic accuracy of severe/complicated hearing loss and/or complicating ear-related conditions in hearing impaired adults. | Month 3
  A physical, "golden standard" ENT assessment was performed control group participants after 3 months. Based on this assessment, participants were again divided into categories of simple hearing loss, severe/complicated hearing loss, and no hearing loss respectively. The "golden standard" ENT assessment at Month 3 was compared to the physical ENT assessment at baseline and diagnostic differences were registered.
  Outcome measures: Sensitivity and specificity of the conventional physical ENT specialist assessment routine in identifying severe/complicated hearing loss and/or complicating ear-related conditions in hearing impaired adults.
Remote vs. physical ENT assessment on correct diagnosis of severe/complicated hearing loss and/or complicating ear-related conditions. | Month 3
  Comparison of sensitivity and specificity of remote vs. physical ENT assessment on correct identification of severe/complicated hearing loss and/or complication ear-related conditions in hearing impaired adults (p-values for comparison).

SECONDARY OUTCOMES:
Patient-reported treatment effect | Month 3
  The Speech, Spatial- and Qualities of Hearing Scale questionnaire af hearing aid treatment (SSQ12B) provides a score correlated to the subjective hearing difficulty severity after hearing aid treatment is initiated.
  Possible scores ranged from -5 (a worsening of conditions after HAs) to 5 (an improvement of conditions after HAs).
Effect of hearing aid treatment | Month 3
  The International Outcome Inventory for Hearing Aids (IOI-HA) covers a minimal set of seven core outcome items. The items are practically oriented and comprise a mini-profile more than a scale.
Patient-reported satisfaction | Month 1
  A validated 21-item questionnaire regarding patient satisfaction during and after project participation was administered.
  The scale ranged from 1-5 (low scores were associated with dissatisfaction, high scores to a high level of satisfaction)
Patient-reported satisfaction | Month 2
  A validated 21-item questionnaire regarding patient satisfaction during and after project participation was administered.
  The scale ranged from 1-5 (low scores were associated with dissatisfaction, high scores to a high level of satisfaction)
Patient-reported satisfaction | Month 3
  A validated 21-item questionnaire regarding patient satisfaction during and after project participation was administered.
  The scale ranged from 1-5 (low scores were associated with dissatisfaction, high scores to a high level of satisfaction)
HA usage time | Month 3
  Overall and average daily usage time (hours) was registered digitally from the hearing aids 3 months after treatment initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Morten Hoegsbro, MD, PhD, MSc, Study Director — Department of Otorhinolaryngology and Audiology, Aalborg University Hospital, Denmark
Locations (1):
- Department of Otorhinolaryngology and Audiology, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Siggaard LD, Jacobsen H, Hougaard DD, Hogsbro M. Digital vs. physical ear-nose-and-throat specialist assessment screening for complicated hearing loss and serious ear disorders in hearing-impaired adults prior to hearing aid treatment: a randomized controlled trial. Front Digit Health. 2023 Jun 8;5:1182421. doi: 10.3389/fdgth.2023.1182421. eCollection 2023. PMID 37363275